CLINICAL TRIAL: NCT04687215
Title: Spinal Cord Stimulation Improves Pain, Arterial Stiffness and Vascular Flow in Lower Extremities in Patients With Diabetes Mellitus Type II A Multidisciplinary Collaborative Prospective Study
Brief Title: Diabetic Neuropathy in Spinal Cord Stimulator Patients
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB20-1098
Record Dates: First submitted 2020-12-09; First posted 2020-12-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus; Neuropathy; Neuropathic Pain; Vascular Diseases; Vascular Stiffness; Microvascular Changes; Pain, Chronic
MeSH Terms: conditions — Diabetes Mellitus; Neuralgia; Vascular Diseases; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients receiving a spinal cord stimulator: Patients that have been seen in the diabetic foot clinic will be evaluated for participation in the study once they have been referred to one of our pain clinics.

SUMMARY:
The objective of this study is to assess the effect Spinal Cord Stimulators have toward improving vascular changes of diabetes mellitus in patients eligible for SCS placement based on their condition of painful diabetic neuropathy; we will evaluate improving their disability and quality of life, improving micro-circulatory changes induced by Diabetes Mellitus (DM), improving macro-circulatory changes induced by DM and improving arterial stiffness of the vessels of the lower extremity.

DETAILED DESCRIPTION:
This is a single-center, pilot study to investigate a preventative modality, spinal cord neuromodulation, that would contribute to reversing the physiologic changes that occur in the lower extremities of diabetic patients. Patients who have been diagnosed with DM type II for at least 1 year and refractory painful diabetic peripheral neuropathy of the lower extremities who are scheduled to receive a spinal cord stimulator may be enrolled in this study pending eligibly for all other criteria.

Once eligibility and consent have been confirmed, each subject will go through a baseline visit where data will collected through a series of questionnaires, a clinical and psychological evaluation by a licensed professional. Subjects will be asked to come back for a series of vascular test prior to their device implantation. This vascular testing will be done at the vascular lab at the University of Chicago Medical Center by trained vascular physicians and techs.

Prior to any study related procedures, all subjects must first sign the approved ICF. This will be performed by the PI or an approved member of the study staff who has been delegated by the PI do so and in a private setting with ample time given to the subject to review and ask any questions regarding the study. Once the ICF has been signed, a copy will be given to the subject and the original will be placed in their research or medical chart.

Background Data

Once the ICF has been complete, demographic data such as name, age, gender will be collected. Along with demographic information, we will collect medical, surgical and medication history for each subject at the initial baseline visit.

Vascular Testing

Before the Spinal Cord Stimulator procedure, all patients enrolled in the study will undergo baseline vascular testing. The following test will be performed on each subject. Subjects will only go through this portion of the study if they receive pre-certification by their insurance for their SCS procedure. Below is a list of tests that will be performed:

1. Flow mediated arterial dilation and by measuring pedal and digital level waveforms and pressure.
2. Doppler flowmetry (Laser Doppler flowmetry if available) by Duplex Scan of lower extremities
3. Ankle Brachial Index
4. Pulse Pressure and aortic pulse wave velocity
5. Peripheral vascular compliance of the lower extremity

   SCS Procedure

   The SCS procedure is being done as part of the subject's clinical care. The subject would be receiving this procedure, even if they do not agree to participate in this study. All patients will have 2 temporary SCS trial leads placed transcutaneously and tunneled to limit the risk for infection. At the end of the trial interval, patients will repeat the vascular testing at 2 weeks post-op at the time just prior to device removal, as well as complete the clinical evaluations as above.

   The SCS waveform used will be consistent and similar for all patients enrolled; at 1 week, study will allow minor SCS waveform modifications to recapture stimulation, but waveforms will be maintained within established parameters in accordance with device used. All patients will attempt to complete the 2 weeks trial; early removal will be performed for the following situations: intolerable pain with stimulation (increase pain >4 points from baseline), infection, neurological deficit (sensory of motor), patient request. Leads will be pulled 2 weeks after placement and patients will be seen 1 week after the leads are pulled. At that time, patient will exit the study and can choose definitive implantation if satisfied with the trial results.

   Study Questionnaires and Assessments

   At various time intervals, all subjects will be asked to complete a series of questionnaires and assessments. These questionnaires are intended to evaluate their quality of life, pain levels, patient satisfaction, functional capacities and mental health. All questionnaires are validated and have been chosen for a specific study endpoint. Below is the list of questionnaires and a brief description of each one. For more specific details on when each will be administered, please refer to the schedule of events (Appendix A).

   List of Questionnaires
   * Numerical Rating Scale (NRS)

     * Assessment for rating pain on a numerical scale
   * Michigan Diabetic Neuropathy Score (MDNS) o Assessment used to assess the degree of diabetic neuropathy
   * Patient Global Impression of Change (PGIC)

     o Used to assess subject satisfaction
   * Oswestry Disability Index (ODI)

     o Used to assess a subject's functional capacity
   * Health Related Quality of Life (H-RQol)

     o Assesses physical and mental health over time
   * Short Form McGill Pain Questionnaire (SF-MPQ)

     o Assesses both the subject's intensity and quality of pain
   * Medication Quantification Scale III (MQS-III) o Used to quantify medication regimen

   Study Visits

   This study consists of 5 total clinic visits. Subjects will be asked to come back prior to their temporary SCS placement for a series of vascular testing. If the subject's insurance does not pre-certify them for the trial SCS procedure, the vascular testing will not be completed and they will be withdrawn from the study. For specific detail in what each visit entails, please refer to the study SCHEMA.

   Below are the list of visits and when they occur.

a. Visit 1 (Baseline) b. Visit 2 (Vascular Testing) c. Visit 3 (1 Week-Post Procedure Visit) d. Visit 4 (2 Weeks-Post Procedure Visit) e. Visit 5 (1 Week Post-Lead Pull Visit)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with DM type 2 of more than 1-year duration
2. DM stage 3 or less
3. Patients ≥18 years of age
4. Refractory painful diabetic peripheral neuropathy of the lower extremities
5. ABI index <0.9

Exclusion Criteria:

1. Patients on anticoagulants
2. Patients with active infections
3. Patients with HbA1>10
4. Psychiatric disorders and cognitive dysfunctions
5. Illicit Drug Usage
6. Patients on dialysis
7. BMI>35.0
8. Surgery within the last 30 days
9. Ulcer of the lower extremities
10. Calcification of the peripheral arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have been seen in the diabetic foot clinic will be evaluated for participation in the study once they have been referred to one of our pain clinics. The study will focus on enrolling patients in early stages of DM 2 with no neuropathic ulcers or arterial calcification.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Improve vascular changes | 6 Weeks
  Improve vascular changes (macroscopic: color, edema, ulceration, etc)
Vascular improvement on lower extremities with the Ankle Brachial Index (ABI) | 6 weeks
  Collect data on possible macrovascular improvement in lower extremities by performing the ABI test
Vascular improvement on lower extremities with the Toe Brachial Index (TBI) | 6 Weeks
  Collect data on possible macrovascular improvement in lower extremities by performing the TBI test
Vascular improvement on lower extremities with the Doppler Flowmetry | 6 Weeks
  Collect data on possible macrovascular improvement in lower extremities by performing the Doppler Flowmetry

SECONDARY OUTCOMES:
Show Improvement in pain in patients with painful diabetic neuropathy | 6 Weeks
  Improve pain in patients with painful diabetic neuropathy by using the Numeric Rating Scale (NRS) that ranges from 0-10 on the pain scale.
Patients' Global Impression of Change (PGIC) | 6 Weeks
  Patient satisfaction using PGIC from baseline to 6 weeks
Health-related quality of life (H-RQol) | 6 Weeks
  Quality of life from baseline to 6 weeks
Oswestry Low Back Pain Disability Questionnaire (ODI) | 6 Weeks
  Functional capacity using the ODI from baseline to 6 weeks
Short-form McGill Pain Questionnaire ( SF-MPQ) | 6 Weeks
  Quality of life
Medication Quantification Scale Version III (MQS-III) | 6 Weeks
  Identify changes in analgesic medication use from 0-6 with the MSQ-III Scale. 0 best outcome and 6 being the worse outcome on the scale
Improve neuropathy markers by using the MICHIGAN DIABETIC NEUROPATHY SCORE (MDNS) | 6 weeks
  Improved Neuropathy in subjects from baseline to 6 weeks by using the MDNS
Improve neuropathy markers by using Clinical Neurological Exam (CNS) | 6 Weeks
  Improve neuropathy markers from baseline to 6 weeks, by using the CNS
Vascular improvement on lower extremities by performing the flow mediated arterial dilation test | 6 Weeks
  Collect data on possible microvascular improvement in lower extremities by performing the flow mediated arterial dilation test

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Anitescu, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No